CLINICAL TRIAL: NCT00290758
Title: Phase IIB Trial of G-2535 (Unconjugated Isoflavones-100) in Women at High Risk for Breast Cancer
Brief Title: Genistein in Preventing Breast Cancer in Women at High Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00840; NCI-2009-00840 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000652922; NCI-04B3 (Other: Northwestern University); NWU03-1-04 (Other: DCP); N01CN35157 (NIH)
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (genistein) (Experimental): Patients receive oral genistein once daily for up to 6 months.
  Interventions: Drug: genistein; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo once daily for up to 6 months.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Drug: genistein — Given orally
  Other Names: CI 75610; genisteol; genisterin; prunetol; sophoricol
  Arms: Arm I (genistein)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I (genistein)

SUMMARY:
This randomized phase II trial is studying how well genistein works in preventing breast cancer in women at high risk for breast cancer. Chemoprevention is the use of certain drugs to keep cancer from forming, growing, or coming back. The use of genistein may prevent breast cancer in women at high risk for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the effect of genistein on the proliferation of breast epithelial cells obtained by fine needle aspiration (FNA), as measured by Ki-67 labeling index, in women who are at high risk for breast cancer.

SECONDARY OBJECTIVE:

I. Determine the effect of this drug on cellular and molecular parameters using epithelial cells obtained by FNA, nipple aspirate fluid, and blood from these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to menopausal status (premenopausal vs postmenopausal) and history of breast cancer (no history of breast cancer vs history of estrogen receptor [ER] positive breast cancer vs history of ER negative breast cancer). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral genistein once daily.

ARM II: Patients receive oral placebo once daily.

In both arms, treatment continues for up to 6 months in the absence of unacceptable toxicity.

After completion of study treatment, patients are followed at 30-37 days.

ELIGIBILITY:
Inclusion Criteria:

* No known soy intolerance
* At increased risk of developing breast cancer in >= 1 previously unaffected breast, as defined by any of the following:

  * Estimated 5-year risk of developing breast cancer using the Gail model, as defined by 1 of the following:

    * Gail score >= 1.66%
    * Gail score >= 0.1% for women age 20-29 years
    * Gail score >= 1.0% for women age 30-39 years
  * Estimated 5-year risk of developing breast cancer using the Claus model:

    * Claus score >= 1.66%
    * Claus score >= 0.1% for women age 20-29 years
    * Claus score >= 1.0% for women age 30-39 years
  * Prior diagnosis of unilateral in situ or invasive breast cancer OR history of atypical hyperplasia, BRCA 1 and/or BRCA 2 positivity
  * History of lobular carcinoma in situ
* No evidence of breast cancer, as determined by a negative mammogram within the past 6 months and a history and physical
* No previously diagnosed breast cancer unless all systemic therapy (including endocrine therapy) was completed at least 1 year ago
* Pre- or postmenopausal
* ECOG performance status 0-1
* Hemoglobin > 10.0 g/dL
* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 1,000/mm^3
* Creatinine < 2.0 mg/dL
* SGPT < 82 U/L
* SGOT < 68 U/L
* Bilirubin < 3 mg/dL* [Note: * Patients with a higher level of bilirubin due to a familial metabolism may be eligible at the discretion of the investigator]
* Life expectancy > 2 years
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* Must be willing to keep a dietary diary
* No venous thrombosis within the past year
* No unrecognized or poorly controlled thyroid disease
* No other cancer within the past 5 years except nonmelanomatous skin cancer or noninvasive cervical cancer
* No other medical condition that, in the opinion of the investigator, would jeopardize either the patient or the integrity of the data obtained
* None of the following for >= 2 weeks before the first random fine needle aspiration and during study participation:

  * Oral contraceptives
  * Soy supplements
  * High soy-containing foods
  * Fish oil supplements
  * Multivitamins
  * Vitamins C and E
  * Daily aspirin or nonsteroidal
  * Anti-inflammatory drugs
* No other concurrent investigational agents
* No concurrent warfarin or other blood thinners
* Female patient

Exclusion Criteria:

Women previously diagnosed with breast cancer will not be eligible unless all systemic therapy (including endocrine therapy) was completed at least one year previously

* Currently pregnant, or planning to become pregnant during the study period
* History of venous thrombosis within past year
* Medical conditions, which, in the opinion of the investigators would jeopardize either the patient or the integrity of the data obtained
* History of other cancer within the past five years, excluding non-melanomatous skin cancer, and non-invasive cervical cancer
* Known soy intolerance
* Unrecognized or uncontrolled thyroid disease, subjects may be on synthroid, but thyroid function must be in normal range or the patient's physician must document that the patient's thyroid is controlled.
* Currently receiving any other investigational agents
* Currently on coumadin, or other blood thinners
* History of breast augmentation implants.
* Rusults from patients who have <4000 epithelial cells in either the first or the second random Fine-needle aspiration (rFNA) will not be included in the study.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan SA, Chatterton RT, Michel N, Bryk M, Lee O, Ivancic D, Heinz R, Zalles CM, Helenowski IB, Jovanovic BD, Franke AA, Bosland MC, Wang J, Hansen NM, Bethke KP, Dew A, Coomes M, Bergan RC. Soy isoflavone supplementation for breast cancer risk reduction: a randomized phase II trial. Cancer Prev Res (Phila). 2012 Feb;5(2):309-19. doi: 10.1158/1940-6207.CAPR-11-0251. PMID 22307566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to accrual January 6, 2006. Study closed to accrual August 27, 2008. Subjects were recruited from the Lynn Sage Comprehensive Breast Center of Northwestern University, through ads on public transportation, through website and flyer distributions.
Pre-assignment Details: Potential subjects underwent a 2 week washout period of soy products, vitamins, and daily aspirin prior to a screening random fine need aspiration (rFNA) of the breast(s). Subjects for which 4,000 or more epithelial cells were obtained the first or second rFNA were considered eligible for study participation.
Groups:
- Arm A (Genistein): Patients received oral genistein once daily for 6 months
- Arm B (Placebo): Patients received oral placebo once daily for 6 months
Period: Pre-Intervention rFNA Through Follow-Up
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Started | 62 | 64
First rFNA Tissue Collection | 62 | 64
Randomization | 62 | 62
Treatment | 61 | 64
Post Intervention Follow-Up | 55 | 54
Completed | 55 | 54
Not Completed | 7 | 10
Not completed — Adverse Event | 1 | 2
Not completed — ConMeds | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Medical Contraindication | 1 | 0
Not completed — Non Compliant | 0 | 1
Period: Post Intervention rFNA
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Started | 55 | 54
Completed | 49 | 49
Not Completed | 6 | 5
Not completed — <4000 Epithelial Cells | 6 | 5

BASELINE CHARACTERISTICS:
Population: Participants who had >4000 epithelial cells in the first and the second rFNA sample.
Groups:
- Arm A: Patients receive oral genistein once daily for up to 6 months.
- Arm B: Patients receive oral placebo once daily for up to 6 months.
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 63 | 124
  >=65 years | 1 | 1 | 2
Gender [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 60 | 62 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 12 | 19
  White | 54 | 52 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Breast Epithelial Cell Proliferation as Measured by Ki-67 Labeling
Description: Breast epithelial tissue samples are used to measure the expression of the cell proliferation marker Ki-67, by counting the percentage of positive MIB-1 immunostained cells, denoted the Ki-67 labeling index. Mean change in the Ki-67 labeling index is assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: Participants who had more than 4,000 epithelial cells in rFNA samples at both baseline and 6 month follow up, met the criteria for compliance, and were available for evaluation of Ki-67 labeling index at both time points. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: Ki-67 labeling index
Groups:
- Arm A (Genistein): Patients receive oral genistein once daily for up to 6 months.
- Arm B (Placebo): Patients receive oral placebo once daily for up to 6 months.
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Number analyzed (Participants) | 49 | 49
Ki-67 labeling index
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 4 | 2
  Postmenopausal with ER- Cancer | .325 (.343) | .289 (.541)
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 2 | 5
  Postmenopausal with ER+ Cancer | -.418 (.191) | -.461 (.458)
  Postmenopausal Without Cancer: number analyzed (Participants) | 14 | 15
  Postmenopausal Without Cancer | -.092 (.525) | -.122 (.735)
  Premonopausal with ER- Cancer: number analyzed (Participants) | 2 | 2
  Premonopausal with ER- Cancer | -.335 (.930) | .873 (.786)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 4 | 4
  Premenopausal with ER+ Cancer | -.387 (.806) | -.204 (1.329)
  Premenopausal without cancer: number analyzed (Participants) | 23 | 21
  Premenopausal without cancer | 1.171 (2.922) | 0.557 (1.546)

2. Secondary Outcome: Measurement of Change in Concentration of Epidermal Growth Factor (EGF) Found in Nipple Aspirate Fluid (NAF)
Description: Mean change in the concentration of EGF found in nipple aspirate fluid is assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: NAF collection was attempted on all 98 participants and was successful in 46 at both time points. Mean change in EGF concentration available for 43 participants. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Number analyzed (Participants) | 23 | 20
ng/ml
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 2 | 0
  Postmenopausal with ER- Cancer | -133.07 (308.28) |
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 0 | 2
  Postmenopausal with ER+ Cancer |  | -197.8 (16.01)
  Postmenopausal without cancer: number analyzed (Participants) | 6 | 5
  Postmenopausal without cancer | 201.05 (380.72) | -38.74 (226.18)
  Premenopausal with ER- Cancer: number analyzed (Participants) | 1 | 2
  Premenopausal with ER- Cancer | -93.23 (0) | 37.38 (69.11)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 0 | 1
  Premenopausal with ER+ Cancer |  | 20.63 (0)
  Premenopausal without cancer: number analyzed (Participants) | 14 | 10
  Premenopausal without cancer | -9.16 (296.55) | -9.26 (175.57)

3. Secondary Outcome: Change in Cytomorphologic Assessment of Atypia and Spectral Imaging Analysis of Atypica Features in Epithelial Cells.
Description: Cytologic atypia evaluation was performed on Papanicolau stained Thin Prep slides using standard criteria, which were also used for spectral spatial imaging. Cell clusters were used to generate image stacks with the Nuance LCTF-based imaging system (CRI Inc). The image data was collected as percent pixels assigned as "atypical". Mean change in the percent pixels assigned "atypical" is assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: Percent pixels
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Number analyzed (Participants) | 49 | 49
Percent pixels
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 4 | 2
  Postmenopausal with ER- Cancer | -1.25 (0.96) | 0 (0)
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 2 | 5
  Postmenopausal with ER+ Cancer | -3.00 (2.12) | -.40 (0.89)
  Postmenopausal Without Cancer: number analyzed (Participants) | 14 | 15
  Postmenopausal Without Cancer | -0.50 (1.87) | 0 (1.45)
  Premenopausal with ER- Cancer: number analyzed (Participants) | 2 | 2
  Premenopausal with ER- Cancer | 0.50 (0.71) | 0 (0)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 4 | 4
  Premenopausal with ER+ Cancer | 0.50 (1.29) | -0.75 (0.96)
  Premenopausal without cancer: number analyzed (Participants) | 23 | 21
  Premenopausal without cancer | 0.17 (2.42) | 0.95 (2.18)

4. Secondary Outcome: Breast Endocrine Environment Measured in Nipple Aspiration Fluid (NAF): Estradiol
Description: Mean change in concentration of estradiol measured in nipple aspiration fluid assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: NAF collection was attempted on all 98 participants and was successful in 46 at both time points. Mean change in estradiol concentration available for 40 participants. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Arm I (Genistein) | Arm II (Placebo)
Number analyzed (Participants) | 21 | 19
pg/ml
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 2 | 0
  Postmenopausal with ER- Cancer | 2251.92 (292.66) |
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 0 | 1
  Postmenopausal with ER+ Cancer |  | -497.3 (0)
  Postmenopausal Without Cancer: number analyzed (Participants) | 5 | 6
  Postmenopausal Without Cancer | -354.39 (643.44) | 925.83 (955.71)
  Premenopausal with ER- Cancer: number analyzed (Participants) | 1 | 2
  Premenopausal with ER- Cancer | -129.58 (0) | -36.38 (16.42)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 0 | 0
  Premenopausal without cancer: number analyzed (Participants) | 13 | 10
  Premenopausal without cancer | -591.81 (992.24) | 6.31 (394.74)

5. Secondary Outcome: Monitor Drug Delivery by Measuring Plasma Genistein by HPLC
Description: Drug delivery is measured be concentration of genistein in plasma using High Performance Liquid Chromatography (HPLC). Mean change in concentration of plasma genistein is assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: Analysis performed by menopause and cancer status.
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Number analyzed (Participants) | 49 | 49
ng/ml
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 4 | 2
  Postmenopausal with ER- Cancer | 368.62 (389.24) | 0 (0)
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 2 | 5
  Postmenopausal with ER+ Cancer | 65.20 (92.20) | 0 (0)
  Postmenopausal Without Cancer: number analyzed (Participants) | 14 | 15
  Postmenopausal Without Cancer | 190.42 (226.17) | 0.65 (2.52)
  Premenopausal with ER- Cancer: number analyzed (Participants) | 2 | 2
  Premenopausal with ER- Cancer | 472.09 (350.16) | 4.56 (6.44)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 4 | 4
  Premenopausal with ER+ Cancer | 423.12 (359.00) | 3.80 (4.40)
  Premenopausal without cancer: number analyzed (Participants) | 23 | 21
  Premenopausal without cancer | 269.88 (250.43) | 3.57 (14.99)

6. Secondary Outcome: Plasma Concentration of Sex Hormone Binding Globulin (SHBG)
Time Frame: 6 months - baseline
Population: Plasma concentration of SHBG was not available for 1 patient in Arm A. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Number analyzed (Participants) | 48 | 49
nmol/L
  Postmenopausal with ER- Cancer: number analyzed (Participants) | 4 | 2
  Postmenopausal with ER- Cancer | 7.39 (28.64) | 22.07 (50.65)
  Postmenopausal with ER+ Cancer: number analyzed (Participants) | 2 | 5
  Postmenopausal with ER+ Cancer | -17.84 (0.55) | -8.12 (13.40)
  Postmenopausal Without Cancer: number analyzed (Participants) | 13 | 15
  Postmenopausal Without Cancer | 3.94 (26.42) | -20.49 (50.03)
  Premenopausal with ER- Cancer: number analyzed (Participants) | 2 | 2
  Premenopausal with ER- Cancer | 15.61 (14.79) | -27.34 (12.13)
  Premenopausal with ER+ Cancer: number analyzed (Participants) | 4 | 4
  Premenopausal with ER+ Cancer | 1.99 (15.26) | -14.79 (17.41)
  Premenopausal without cancer: number analyzed (Participants) | 23 | 21
  Premenopausal without cancer | -11.18 (39.90) | 3.79 (29.96)

7. Secondary Outcome: Breast Endocrine Environment Measured in Nipple Aspiration Fluid (NAF): Cathepsin D
Description: Mean change in concentration of Cathepsin D measured in nipple aspiration fluid assessed from baseline to 6 month follow up.
Time Frame: 6 months - baseline
Population: NAF collection was attempted on all 98 participants and was successful in 46 at both time points. Mean change in Cathespin D concentration available for 44 participants. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: mg/ml
Arm/Group | Arm I (Genistein) | Arm II (Placebo)
Number analyzed (Participants) | 23 | 21
mg/ml
  post menopausal with ER- cancer: number analyzed (Participants) | 2 | 0
  post menopausal with ER- cancer | -3105.29 (6764.20) |
  post menopasual with ER+ caner: number analyzed (Participants) | 0 | 2
  post menopasual with ER+ caner |  | -3961.16 (1295.29)
  post menopausal without cancer: number analyzed (Participants) | 6 | 5
  post menopausal without cancer | 3362.326 (9545.02) | -1774.72 (17644.27)
  pre menopausal with ER- cancer: number analyzed (Participants) | 1 | 2
  pre menopausal with ER- cancer | 1800.40 (0) | 29337.79 (36645.39)
  pre menopausal with ER+ cancer: number analyzed (Participants) | 0 | 1
  pre menopausal with ER+ cancer |  | -6218.25 (0)
  Pre menopausal without Cancer: number analyzed (Participants) | 14 | 11
  Pre menopausal without Cancer | -4904.09 (28128.12) | 486.56 (40420.50)

8. Secondary Outcome: Breast Endocrine Environment Measured in Nipple Aspiration Fluid (NAF): ps2
Description: Mean change in concentration of protein ps2 measured in nipple aspiration fluid assessed from baseline to 6 month follow up.
Time Frame: 6 month - baseline
Population: NAF collection was attempted on all 98 participants and was successful in 46 at both time points. Mean change in ps2 concentration available for 44 participants. Analysis performed by menopause and cancer status.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm I (Genistein) | Arm II (Placebo)
Number analyzed (Participants) | 23 | 21
ng/ml
  Post menopausal with ER- cancer: number analyzed (Participants) | 2 | 0
  Post menopausal with ER- cancer | -28.00 (41.85) |
  Post menopasual with ER+ caner: number analyzed (Participants) | 0 | 2
  Post menopasual with ER+ caner |  | -61.06 (10.06)
  Post menopausal without cancer: number analyzed (Participants) | 6 | 5
  Post menopausal without cancer | -14.17 (32.40) | -6.10 (65.38)
  Pre menopausal with ER- cancer: number analyzed (Participants) | 1 | 2
  Pre menopausal with ER- cancer | -16.68 (0) | 4.69 (23.75)
  Pre menopausal with ER+ cancer: number analyzed (Participants) | 0 | 1
  Pre menopausal with ER+ cancer |  | -31.46 (0)
  Pre menopausal without Cancer: number analyzed (Participants) | 14 | 11
  Pre menopausal without Cancer | -20.49 (54.30) | 12.17 (29.74)

ADVERSE EVENTS:
Time Frame: 3 years
Description: February, 2006 th March, 2009
Groups:
- Arm A (Genistein): Patients take oral genistein once daily for up to 6 months.
- Arm B (Placebo): Patients take oral placebo once daily for up to 6 months.
Arm/Group | Arm A (Genistein) | Arm B (Placebo)
Serious Adverse Events (participants affected / at risk) | 6/62 | 1/64
Other Adverse Events (participants affected / at risk) | 50/62 | 56/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genistein) (N=62) | Arm B (Placebo) (N=64)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mood Alteration: Depression (Nervous system disorders) | 1 (1) | 0 (0)
renal - Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstruction, GU: Uterus (Renal and urinary disorders) | 1 (1) | 0 (0)
Sexual (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory: Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Genistein) (N=62) | Arm B (Placebo) (N=64)
Hemorrhage - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Bloody Nipple Discharge
Hemorrhage with Surgery (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood/bone marrow: Blood- Other (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Anemia
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytes (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Edima: Limb (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Coagulation - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Coagulopathy
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Arrythmia - Select Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardia Ischemia/Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Inner Ear Infection
Hot Flashes (Endocrine disorders) | 10 (11) | 8 (10)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Endocrine - Other (Endocrine disorders) | 1 (2) | 0 (0) — Night Sweats
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Other (Eye disorders) | 1 (1) | 0 (0) — Blurred Vision
Ocular - Other (Eye disorders) | 0 (0) | 2 (4) — BILATERAL EYE ITCHING/IRRITATION
Flashing Lights (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 5 (6)
nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Heartburn (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
GI - Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Colon Polyps
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain - Other (General disorders) | 2 (2) | 0 (0) — Axillary Soreness
Pain - Select: Throat/Pharynx/Larynx (General disorders) | 3 (3) | 4 (5)
Pain - Select: Larynx (General disorders) | 0 (0) | 1 (1)
Pain - Select: Back (General disorders) | 4 (7) | 3 (5)
Pain - Select: Joint (General disorders) | 3 (6) | 6 (7)
Pain - Select: Breast (General disorders) | 4 (5) | 5 (5)
Pain - Select: Extremity - Limb (General disorders) | 1 (2) | 4 (5)
Pain - Select: Head/Headaches (General disorders) | 6 (9) | 6 (6)
Pain - Select: Cardiac/Heart (General disorders) | 0 (0) | 1 (1)
Pain - Select: Abdomen Nos (General disorders) | 2 (2) | 0 (0)
Pain - Select: Neuralgia (General disorders) | 0 (0) | 1 (1)
Pain - Select: Eye (General disorders) | 0 (0) | 1 (1)
Pain - Select: Bone (General disorders) | 0 (0) | 1 (2)
Pain - Select: Skin (General disorders) | 2 (4) | 0 (0)
Pain - Select: Uterus (General disorders) | 2 (2) | 0 (0)
Pain - Select: Dental/Teeth/Peridontal (General disorders) | 0 (0) | 1 (1)
Constitutional Symptoms - Other (General disorders) | 3 (3) | 4 (5) — Malaise
Constitutional Symptoms - Weight Gain (General disorders) | 2 (2) | 0 (0)
Constitutional Symptoms - Fever (General disorders) | 10 (10) | 2 (2)
Constitutional Symptoms - Fatigue (General disorders) | 1 (1) | 3 (4)
Constitutional Symptoms - Insomnia (General disorders) | 3 (3) | 2 (2)
Constitutional Symptoms - Rigors/Chills (General disorders) | 1 (1) | 0 (0)
Constitutional Symptoms - Sweating (General disorders) | 0 (0) | 1 (1)
Allergic Reastion (Immune system disorders) | 0 (0) | 1 (6)
Infection (documented clinically) Select: Bladder (Urinary) (Infections and infestations) | 0 (0) | 1 (1)
Infection with Unknown ANC - Select: Bronchus (Infections and infestations) | 2 (2) | 1 (1)
Infections - Other (Infections and infestations) | 3 (3) | 5 (5) — Sinus Infection
Infection with Unknwn ANC - Select: Vagina (Infections and infestations) | 3 (3) | 2 (4)
Infection with Unknown ANC - Select: Skin (Cellulitis) (Infections and infestations) | 1 (1) | 0 (0)
Infection (Documented ClinicallY) - Select: Vagina (Infections and infestations) | 1 (1) | 0 (0)
Infection With Unknown ANC - Select: Upper Airways Nose (Infections and infestations) | 0 (0) | 1 (2)
Infection With Unknown ANC - Select: Sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection With Unknown ANC - Select: Urinary Tract Nos (Infections and infestations) | 0 (0) | 2 (2)
Infection (Documented Clinically) - Select: Sinus (Infections and infestations) | 0 (0) | 1 (1)
Infection With Unknown ANC - Select: Conjunctiva (Infections and infestations) | 0 (0) | 1 (1)
Infection (Documented Clinically) - Select: Urinary Tract Nos (Infections and infestations) | 0 (0) | 1 (1)
Infection (Documented Clinically) - Select: Pleura (Empyema) (Infections and infestations) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ALt (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
AST (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cholesterol (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal - Other (Specify) (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (7) — Right Lateral Side Discomfort
Joint - Function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mood Alteration - Select: Anxiety (Nervous system disorders) | 4 (4) | 2 (2)
Mood Alteration - Select: Depression (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Neurology (Other) (Nervous system disorders) | 1 (1) | 0 (0) — NUMBNESS, TINGLING, PAIN LEFT UPPER ARM
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Incontinence, Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstruction, GU - Select:: Uterus (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal - Other (Renal and urinary disorders) | 2 (2) | 1 (1) — vaginal itching
Urinary Frequesncy (Renal and urinary disorders) | 1 (1) | 0 (0)
Sexual - Other (Reproductive system and breast disorders) | 6 (6) | 8 (12) — MENORRHAGIA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 10 (16)
Pulmonary - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 0 (0) — Sneezing
Pulmonary/Upper Respiratory - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 15 (23) — Sinus Congestion
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (4) — MOLE REMOVED ON ABDOMEN - SHOWED DYSPLASIA
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Wound Compilation - Non-Infectious (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less